CLINICAL TRIAL: NCT03490825
Title: Enhancing Circadian Signal to Improve Cardiometabolic Function in Aging
Brief Title: Aging Program Project Grant 6
Acronym: PPG6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Phyllis Zee, Professor of Neurology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STU00206014
Record Dates: First submitted 2018-03-30; First posted 2018-04-06 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2024-03

CONDITIONS: Improving Cardiometabolic Outcomes in Older Adults
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: The study is designed as a randomized controlled trial where each participant will receive one of four intervention types. Subjects will be randomized at baseline visit to one of four arms using a randomized block design to achieve balanced groups. Randomization will be stratified by sex. The allocation will be created using an online randomization tool. This study will include a 6 week four arm field intervention to evaluate the independent effect of meal timing or melatonin as well as their combined effects
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Meal timing + Melatonin (Experimental): This arm will consist of imposing a minimum overnight fasting period of 12 hours and a maximum of 16 hours (with exception of water and other non-caloric beverages), beginning 3 hours before their habitual bed time. This arm will also include a 1mg melatonin supplementation given daily during the intervention.
  Interventions: Dietary Supplement: Melatonin 1 mg; Other: Meal timing
- Meal timing + Placebo (Experimental): This arm will consist of imposing a minimum overnight fasting period of 12 hours and a maximum of 16 hours (with exception of water and other non-caloric beverages), beginning 3 hours before their habitual bed time. This arm will also include a melatonin placebo (Lactose/Starch) supplementation given daily during the intervention.
  Interventions: Dietary Supplement: Placebos; Other: Meal timing
- Melatonin (Experimental): This arm will continue to eat at their habitual meal times, and maintain their average habitual caloric and macronutrient intake. No EOF will be imposed. This arm will include a 1mg melatonin supplementation given daily during the intervention.
  Interventions: Dietary Supplement: Melatonin 1 mg; Other: Non-Meal timing
- Placebo (Placebo Comparator): This arm will continue to eat at their habitual meal times, and maintain their average habitual caloric and macronutrient intake. No EOF will be imposed. This arm will also include a melatonin placebo (Lactose/Starch) supplementation given daily during the intervention.
  Interventions: Dietary Supplement: Placebos; Other: Non-Meal timing

INTERVENTIONS:
Dietary Supplement: Melatonin 1 mg — Melatonin (1mg) will be administered daily during the intervention. Melatonin capsules will be obtained from Life Extension (Ft. Lauderdale, FL). The investigational drug pharmacy (IDP) at Northwestern Memorial Hospital will encapsulate the melatonin pills so the placebo (lactose) and melatonin pills appear identical. We have worked with this IDP on other projects. The investigators on this study have experience in administering melatonin for investigational and clinical purposes.
  Arms: Meal timing + Melatonin; Melatonin
Dietary Supplement: Placebos — Placebo will be administered daily during the intervention. The investigational drug pharmacy (IDP) at Northwestern Memorial Hospital will encapsulate the pills so the placebo (lactose/starch) and melatonin pills appear identical. We have worked with this IDP on other projects. The investigators on this study have experience in administering melatonin for investigational and clinical purposes.
  Arms: Meal timing + Placebo; Placebo
Other: Meal timing — Subjects are instructed to maintain an extended overnight fasting period of 12-16 hours.
  Other Names: Extended overnight fasting (EOF)
  Arms: Meal timing + Melatonin; Meal timing + Placebo
Other: Non-Meal timing — Subjects are instructed to maintain their habitual meal timing.
  Other Names: Non-extended overnight fasting (nEOF)
  Arms: Melatonin; Placebo

SUMMARY:
This study aims to enhance circadian signals to improve cardiometabolic functions in older adults though meal timing interventions and melatonin supplements. Cardiometabolic disease (CMD) is prevalent among older adults, but despite vigorous research to prevent it, it remains on of the greatest public health challenges. Previous research has shown that extended overnight fasting and melatonin supplements may enhance circadian signals which in turn would enhance cardiometabolic function in older adults.

This study will place subjects in one of four intervention groups, 1) Meal timing + Melatonin, 2) Meal timing + Placebo, 3) Melatonin, or 4) Placebo in order test out the effects of meal timing and melatonin both separately and together and cardio metabolic functions. The study will explore the effects of these interventions in acute-based setting and extended-based settings. This will allow us to test out the hypotheses of the study that meal timing can improve amplitude of circadian signals and improve cardiometabolic functions and sleep quality as well as melatonin improving cardiometabolic function and sleep quality. Finally, we will determine if the the addition of melatonin will further enhance the effects of the meal timing intervention for improving cardiometabolic function and sleep.

ELIGIBILITY:
Inclusion Criteria:

* Older adults 55-75 years old.
* Females must be post-menopausal.
* BMI 25-45
* Regular eating schedule (consuming at least 2 meals/day) and sleeping schedules (deviation of ≤ 2 hours in daily mid-sleep time).
* Self-report sleep duration of ≥ 6.5 hours.
* Habitual mid-sleep time of 1-5 am.
* Habitual time in bed less than 9 hours
* HbA1c <6.5
* Habitual overnight fast of ≤ 13 hour (Determined by a mean overnight fast ≤ 13 hours over 3 days of self-monitoring of food intake)

Exclusion Criteria:

* History or current diagnosis of a primary sleep disorder (Chronic insomnia, restless leg syndrome, parasomnias, sleep apnea).
* AHI ≥30
* History of anemia.
* Diagnosis of diabetes or currently on any medications for diabetes.
* Endocrine dysfunction including PCOS.
* History of cognitive or other neurological disorders.
* History of DSM-V criteria for any major psychiatric disorder.
* Beck depression Index (BDI) of ≥16 indicating moderate depression.
* Mini mental status Exam <26 indicating cognitive impairment.
* Unstable or serious medical conditions.
* Individuals with pacemakers, defibrillators, mediation pumps, or any other implanted device.
* Any GI disease that requires dietary adjustment.
* Current or use within last month of melatonin.
* Current use of psychoactive, hypnotic, stimulants, or pain medications.
* Current use of hormone replacement therapy.
* Shift work or other self-imposed irregular sleep schedules.
* History of habitual smoking (≥6 cigarettes/week).
* Caffeine consumption >400 mg/day.
* Medically managed or self-reported weight loss program within past 6 months.
* Bariatric weight loss surgery.
* Blindness or visual impairment other than glasses.
* Allergic to heparin.
* Adults unable to consent will be excluded.
* Pregnant women will be excluded.
* Prisoners will be excluded.
* Individuals who are not yet adults (infants, children, teenagers) will be excluded.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Matsuda Index | 8 weeks
  The matsuda index of whole body index sensitivity will be calculated to explore the effect of sleep and circadian rhythms on the relationship between EOF, melatonin, and CMD.
Nocturnal Blood Pressure Dipping | 8 weeks
  Defined as a ratio of sleep blood pressure to wake blood pressure less than 0.90.
Melatonin Amplitude | 8 weeks
  The melatonin amplitude will be calculated to determine the effects of the interventions on sleep and CMD outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Zee, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided